CLINICAL TRIAL: NCT06375200
Title: Healthcare for Men with Suicidal Thoughts: Needs Assessment
Acronym: KUJK2NEEDS
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0066
Record Dates: First submitted 2024-04-08; First posted 2024-04-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Suicide Prevention; Help-Seeking Behavior; Men
MeSH Terms: conditions — Suicide Prevention; Help-Seeking Behavior; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Individuals with suicidal thoughts (Questionnaire): Anticipated n=274
  * Adults (≥18y/o)
  * Experienced suicidal thoughts in the past three year
  * Access to internet administered a one time online questionnaire (15-20 min.)
  Interventions: Other: No intervention
- Individuals with suicidal thoughts (Focus Group): Anticipated n=60
  * Adults (≥18y/o)
  * Experienced suicidal thoughts in the past three year
  * Access to internet administered a one time online background questionnaire (5-10min.) and partake in a focus group (2h)
  Interventions: Other: No intervention
- Healthcare providers (Questionnaire): Anticipated n=360
  * Healthcare providers (eg GP's, psychiatrists, medical doctors, psychologists, psychotherapists, and nurses working in healthcare) (≥18y/o)
  * Previously encountered men with suicidal thoughts and/or behaviour professionally administered a one time online questionnaire (10-15 min.)
  Interventions: Other: No intervention
- Healthcare providers (Focus group): Anticipated n=20
  * Healthcare providers (eg GP's, psychiatrists, medical doctors, psychologists, psychotherapists, and nurses working in healthcare) (≥18y/o)
  * Previously encountered men with suicidal thoughts and/or behaviour professionally administered a one time online questionnaire (10-15 min.) and optionally partake in an online focus group (2h)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational one-time questionnaire study without intervention

SUMMARY:
The aim of the current project is twofold, namely

1. To gain insight into needs related to help-seeking among men with (previous) suicidal thoughts (STUDY 1). More specifically, this study examines help-seeking behaviour, possible barriers to seeking help and needs with regard to existing tools and health care among men who had suicidal thoughts. In other words, is there a difference in help-seeking behaviour between men and women with suicidal thoughts in the past and what factors contribute to this difference? More specifically:

   1. To what extent do men with suicidal thoughts in the past recognize their need for help, compared to women with suicidal thoughts in the past?
   2. What barriers and needs do men with suicidal thoughts in the past experience towards seeking help, compared to women with suicidal thoughts in the past?
   3. What barriers and needs do men with suicidal thoughts in the past experience to remain engaged in help, compared to women with suicidal thoughts in the past?
2. To map out needs of healthcare providers in working with men with suicidal thoughts and/or behaviour (STUDY 2). More specifically, how do healthcare providers experience working with men who are feeling suicidal and what are their experienced barriers and needs. Two main research questions were formulated:

   1. How do health care providers experience working with men (in comparison to women or people of other genders) who are feeling suicidal?
   2. What needs and barriers do health care providers experience when working with men (in comparison to women or people of other genders) who are feeling suicidal?

DETAILED DESCRIPTION:
Approximately three out of four people who die by suicide are men. Suicide is a complex phenomenon, which cannot be explained by a single factor, but rather is a result of a variety of neurobiological, psychological and social risk factors. Considering the difference in suicide risk between men and women, researchers have tried to identify risk factors specific to men, which might contribute to the increased suicide risk. Differences in help-seeking behaviour and received help have repeatedly been put forward as being one of these factors as men are less likely to seek help and have a higher drop-out rate once having started interventions. That is why in our new project we want to investigate what barriers and needs men experience with regard to existing healthcare and how healthcare can meet these needs.

This will be done in two studies among 1) people with suicidal thoughts in the past 3 years and 2) healthcare providers.

* STUDY 1: A needs assessment among men with a history of suicidal thoughts, consisting of

  * One online needs assessment questionnaire (15-20 min.) for men, women and individuals with other gender identities (≥18y/o) who have experienced suicidal thoughts in the past three years. The questionnaire assesses help-seeking behaviour and factors that may be associated with it (i.e. barriers to help, perceived stigma, emotional openness, self-reliance, perceived need for help, needs regarding healthcare). This questionnaire will be administered to men as well as to women/people with a different gender identity in order to compare the different gender groups.
  * Six online focus groups with men, women and individuals with other gender identities (separately) (≥18y/o) who have experienced suicidal thoughts in the past three years.
* STUDY 2: A needs assessment among healthcare providers, consisting of

  * One online needs assessment questionnaire (10-15 min.) for health care providers (i.e., general practitioners (GP's), psychiatrists, medical doctors, psychologists, psychotherapists and nurses working in healthcare) (≥18y/o) who have previously encountered men with suicidal thoughts and/or behaviour professionally. The questionnaire is used to identify their needs regarding working with men with suicidal thoughts.
  * Two online focus groups with health care provides (GP's, psychiatrists, medical doctors, psychologists, psychotherapists and nurses working in healthcare) (≥18y/o) who have previously encountered men with suicidal thoughts and/or behaviour professionally to further discuss these needs.

ELIGIBILITY:
STUDY 1:

Inclusion Criteria:

* Adults (≥18y/o)
* Experienced suicidal thoughts in the past three year
* Access to internet

Exclusion Criteria:

/

STUDY 2:

Inclusion Criteria:

* Healthcare providers (eg GP's, psychiatrists, medical doctors, psychologists, psychotherapists, and nurses working in healthcare) (≥18y/o)
* Previously encountered men with suicidal thoughts and/or behaviour professionally

Exclusion Criteria:

/

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STUDY 1: adults with suicidal ideation in the past 3 years STUDY 2: healthcare providers working with men with suicidal ideation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
STUDY 1: Help-seeking behavior | Baseline. Completing the questionnaire will take about 15-20 minutes
  Actual help-seeking questionnaire (Rickwood ea, 2005); adapted based on study Tang ea 2023. 9 items to be rated if consulted [yes/no/not applicable] for suicidal thoughts and satisfaction with received support/advice [very dissatisfied, rather dissatisfied, neutral, rather satisfied, very satisfied]
STUDY 1: Experienced need | Baseline. Completing the questionnaire will take about 15-20 minutes
  Single item from study Tang et al., 2022 [on a scale from 0-10]
STUDY 1: Emotional Openness | Baseline. Completing the questionnaire will take about 15-20 minutes
  Self-developed question need/possibility for openness about suicidal thoughts [no need; insufficient opportunity; moderate opportunity; sufficient opportunity; more than sufficient opportunity] 12-item Distress Disclosure Index (Kahn & Hessling, 2001): 12 items to be rated on a 5-point Likert scale [strongly disagree to strongly agree]
STUDY 1: Barriers | Baseline. Completing the questionnaire will take about 15-20 minutes
  Barriers to Access to Care Evaluation (BACE; Clement ea, 2012): 30 items to be rated on a 4-point Likert scale ([not at al, a little, quite a lot, a lot]
STUDY 1: Self-reliance | Baseline. Completing the questionnaire will take about 15-20 minutes
  CMNI self-reliance factor (Mahalik ea, 2003; Levant ea, 2020): 5 items to be rated on a 4-point Likert scale [strongly disagree, disagree, agree, strongly agree]
STUDY 1: Stigma | Baseline. Completing the questionnaire will take about 15-20 minutes
  Self Stigma Scale for Seeking Help (Vogel ea 2006): 10 items to be rated on a 5-point Likert scale [strongly disagree to strongly agree]
STUDY 1: needs of individuals with suicidal ideation | Baseline. Completing the questionnaire will take about 15-20 minutes
  Needs: 13 needs which they can indicate whether they didn't/don't need, need(ed) but didn't receive or need(ed) and receive(d). Follow-up questions on needed information, needed professional support and needed social contact.
STUDY 2: needs of healthcare providers | Baseline. Completing the questionnaire will take about 10-15 minutes
  self-developed questionnaire: experienced differences in working with men/women with suicidal thoughts [open question; 1 item on general differences on 5-point likert scale; 15 statements of aspects of care with 5-point scale to indicate differences]; needed support in working with suicidal men [open]; need for training [yes/no]; preferred format for training [webinar, e-learning, folder, information on website, study day, physical class, other]; maximum time to be invested in training [<15 minutes, 15-30 minutes, 30 minutes - 1 hour; 1-2 hours; half a day; an entire day; multiple days]; needed information [open]; conditions to partake in training [open]; where do healthcare providers expect to find information on this subject [suicide prevention websites, websites of professional associations, other]; other needs [open]; knowledge of existing tools, trainings and websites [yes/no]; use of existing websites [yes/no]

OTHER OUTCOMES:
STUDY 1: Socio-demographic characteristics | Baseline. Completing the questionnaire will take about 5-10 minutes
  Self-developed: gender [male, female, non-binary, other], age [open], sexual orientation [heterosexual, homosexual, bisexual, asexual, other, prefer not to say, don't know], relationship status [single, in relationship, married/cohabitant, separated, divorced, widowed], location[province and urban/rural], cultural background [Belgian background, Western migration background, non-Western migration background, other], living situation [alone, with partner, with children, with parents, with others, other - multiple options possible], education [no degree, primary education, secondary education, higher education non-university, higher education university] and employment status [student, mainly employed, mainly self-employed, mainly houseman/wife; looking for work, incapacitated, retired].
STUDY 1: Suicidality | Baseline. Completing the questionnaire will take about 15-20 minutes
  Based on Gezondheidenquete 2018: suicidal ideation ever, in the past 12 months and current [yes/no]; suicide attempt ever [1/more than 1/no], in the past 12months
STUDY 2: socio-demographic variables | Baseline. Completing the questionnaire will take about 10-15 minutes
  Self-developed questionnaire: gender [male, female, non-binary, other], age [open], job [GP, psychiatrist, psychologist, psychotherapist, social worker, pedagogue, psychosocial prevention advisor, nurse, other], additional psychotherapy education [yes/no], current employment [private practice, group practice, 'center for general wellbeing', 'center for mental health', psychiatric hospital, psychiatric department of a general hospital, psychiatric center, company, other], location of current employment [province], work experience [<2 years, 2-5 years, 5-10 years, 10-20 years, >20 years]
STUDY 2: Professional experience with men with suicidal thoughts | Baseline. Completing the questionnaire will take about 10-15 minutes
  Professional experience with men with suicidal thoughts [never/rarely, a few times a year, monthly, weekly, daily], subjective experience [very inexperienced, rather inexperienced, a little inexperienced, rather experienced, very experienced], previous suicide attempt of a male patient [yes/no], previous passing a a male patient due to suicide [yes/no]; age group given care to [toddlers and preschoolers, children 6+, youth 14+, adults, elderly 65+ - multiple options possible], format of care provided [individual conversation, family conversation, group conversation; medication; psychotherapeutic support, psychosocial support - multiple options possible]; settings of provided care [work, school, leisure, healthcare, other - multiple options possible]

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang S, Reily NM, Arena AF, Batterham PJ, Calear AL, Carter GL, Mackinnon AJ, Christensen H. People Who Die by Suicide Without Receiving Mental Health Services: A Systematic Review. Front Public Health. 2022 Jan 18;9:736948. doi: 10.3389/fpubh.2021.736948. eCollection 2021. PMID 35118036
- [Background] Stiawa M, Muller-Stierlin A, Staiger T, Kilian R, Becker T, Gundel H, Beschoner P, Grinschgl A, Frasch K, Schmauss M, Panzirsch M, Mayer L, Sittenberger E, Krumm S. Mental health professionals view about the impact of male gender for the treatment of men with depression - a qualitative study. BMC Psychiatry. 2020 Jun 3;20(1):276. doi: 10.1186/s12888-020-02686-x. PMID 32493263
- [Background] Clement S, Brohan E, Jeffery D, Henderson C, Hatch SL, Thornicroft G. Development and psychometric properties the Barriers to Access to Care Evaluation scale (BACE) related to people with mental ill health. BMC Psychiatry. 2012 Jun 20;12:36. doi: 10.1186/1471-244X-12-36. PMID 22546012
- [Background] Kahn JH and Hessling RM (2001) 'Measuring the tendency to conceal versus disclose psychological distress'. Journal of Social and Clinical Psychology, 20(1): 41-65
- [Background] Levant RF, McDermott R, Parent MC, Alshabani N, Mahalik JR, Hammer JH. Development and evaluation of a new short form of the Conformity to Masculine Norms Inventory (CMNI-30). J Couns Psychol. 2020 Oct;67(5):622-636. doi: 10.1037/cou0000414. Epub 2020 Feb 3. PMID 32011153
- [Background] Mahalik, J. R., Locke, B. D., Ludlow, L. H., Diemer, M. A., Scott, R. P. J., Gottfried, M., & Freitas, G. (2003). Development of the Conformity to Masculine Norms Inventory. Psychology of Men & Masculinity, 4(1), 3-25. https://doi.org/10.1037/1524-9220.4.1.3
- [Background] Kwon M, Lawn S, Kaine C. Understanding Men's Engagement and Disengagement When Seeking Support for Mental Health. Am J Mens Health. 2023 Mar-Apr;17(2):15579883231157971. doi: 10.1177/15579883231157971. PMID 36880329
- [Background] Vogel, D. L., Wade, N. G., & Haake, S. (2006). Measuring the self-stigma associated with seeking psychological help. Journal of Counseling Psychology, 53(3), 325-337. https://doi.org/10.1037/0022-0167.53.3.325
- [Background] Rickwood, D., Deane, F. P., Wilson, C. J., & Ciarrochi, J. (2005). Young people's help-seeking for mental health problems. Australian E-Journal for the Advancement of Mental Health, 4(3), 218-251. https://doi.org/10.5172/jamh.4.3.218
- [Background] Tang, S., Reily, N. M., Batterham, P. J., Draper, B., Shand, F., Han, J., Aadam, B., & Christensen, H. (2023). Correlates of non-receipt of formal mental health services among Australian men experiencing thoughts of suicide. Journal of Affective Disorders Reports, 11, 100455. https://doi.org/10.1016/j.jadr.2022.100455